CLINICAL TRIAL: NCT06692777
Title: Evaluation of the Hypolipidemic Effect of Bergavit by a Human Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, You-Cheng Shen, Associate Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS2-22083
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bergavit (Experimental): Group Bergavit : 60 subjects treated with Bergavit capsule intake of 150 mg/die of pure flavonoids for 4 months.
  Interventions: Dietary Supplement: Bergavit
- Placebo (Placebo Comparator): Group Placebo: 60 subjects will take capsule equivalent amount of maltodextrin for 4 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bergavit — Subjects treated with Bergavit capsule intake of 150 mg/die of pure flavonoids for 4 months.
  Arms: Bergavit
Dietary Supplement: Placebo — Subjects will take capsule equivalent amount of maltodextrin for 4 months.
  Arms: Placebo

SUMMARY:
Bergavit is a product contains bergamot. Bergamot is an endemic plant of the Calabrian region in southern Italy with a unique profile of flavonoids and flavonoid glycosides present in its juice and albedo, its flavonoids was able to reduce serum levels of lipids and ameliorate the thickening of the arteries through modulating enzymatic activities, anti-oxidation, anti-inflammatory mechanisms and inhibition of monocyte activation and proliferation.The primary outcome of the study the assessment of the the hypolipidemic effect of Bergavit. The secondary outcomes are the assessment of: a) the hypoglycemic effect of Bergavit, b) the activity of Bergavit on weight loss, and c) the hepatoprotective activity of Bergavit.

DETAILED DESCRIPTION:
The study duration is 4 months. Subjects will attend clinic visits as follows:

* T0: First visit: assessment of all baseline parameters, Beginning of treatment
* T2: Second visit: assessment only of LDL level, Total cholesterol, ox-LDL, Triglycerides level, fasting glucose.
* T3: Third visit: assessment of all parameters.
* T4: Fourth visit: assessment of all parameters, end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1 Healthy men and women (40-70 years old);
* 2 Asian subjects with LDL-cholesterol (ranging from 100 to 159; see here below)
* 3 Subjects naïve to statins or other treatment and food supplement that can interfere with the study treatment for the previous 1 month
* 4 Reading, understanding and signed approval of the informative consent
* 5 No vegetarian. Subjects who will continue, expect reserve, their normal lifestyle
* 6 Healthy volunteers without clinical illness diagnosed with relevant effect on the gastrointestinal system or the motility visceral

Exclusion Criteria:

* 1 Subjects <40 and >70 years old
* 2 Clinical history with relevant presence of any disorder or administration of drugs/food supplement that can potentially interfere with the treatment under study
* 3 lack of compliance defined as not using the correct Bergavit dose or placebo for>1 week), and inability to give informed consent
* 4 Subjects who have changed their diet significantly or have been placed on weight reduction products
* 5 Smokers, Obesity subjects, during breast feeding
* 6 Changing the eating habits within the 2 weeks previous the screening
* 7 During the pregnancy of the subjects or of the subjective planning of the study
* 8 Subjects with a history of drug, alcohol and other substance abuse
* 9 Known food intolerance or food allergy
* 10 Subjects involved in a clinical or food study within the previous month
* 11 Subjects who have unstable medical diseases (cardiac arrhythmias or ischemia, uncontrolled hypertension and hypotension, diabetes mellitus, kidney failure)
* 12 Subjects with a history of paralysis or cerebral vascular accident
* 13 Subjects with active cancers or on chemotherapy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-10-21 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
The Changes of LDL-C of the Subjects. | 16 weeks
  A randomized-double blind trial. The values change of LDL-C between before to after 0, 8, 12, 10 & 16 weeks.

SECONDARY OUTCOMES:
The changes of Cholesterol of the Subjects. | 16 weeks
  A randomized-double blind trial. The values change of Cholesterol between before to after 0, 8, 12, 10 & 16 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan